CLINICAL TRIAL: NCT01380444
Title: A Multi-Center Randomized Controlled Trial of Intramedullary Nails Versus Sliding Hip Screws in the Management of Intertrochanteric Fractures of the Hip
Brief Title: Intramedullary Nail Versus Sliding Hip Screw Inter-Trochanteric Evaluation
Acronym: INSITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: Global Research Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14032012_INSITE_v2.0; 96308751 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Femoral Neck Fractures; Intertrochanteric Fracture
Keywords: Intertrochanteric fracture; Gamma3 intramedullary nail; Sliding hip screw
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- 1 (Active Comparator): Gamma3 Intramedullary Nails
  Interventions: Procedure: Gamma3 Intramedullary Nails (Stryker)
- 2 (Active Comparator): Sliding Hip Screws
  Interventions: Procedure: Sliding Hip Screws

INTERVENTIONS:
Procedure: Gamma3 Intramedullary Nails (Stryker) — The Gamma3 nail is cannulated for Guide-Wire-controlled insertion, and features a conical tip for optimal alignment with the inner part of the cortical bone. A single distal Locking Screw is provided to stabilize the nail in the medullary canal and to help to prevent rotation in complex fractures.
  Other Names: Gamma Nail; Gamma3 Nail; Intramedullary Nail (IM Nail)
  Arms: 1
Procedure: Sliding Hip Screws — The sliding hip screw is a single larger diameter partially threaded screw, which is affixed to the proximal femur with a side plate (with a minimum of two holes and a maximum of four holes) and no supplemental fixation.
  Other Names: Sliding Hip Screw (SHS); Dynamic Hip Screw (DHS); Compression Screw and Side Plate
  Arms: 2

SUMMARY:
The purpose of this study is to assess the impact of Gamma3 intramedullary nails versus sliding hip screws on health-related quality of life as measured by the EuroQuol-5D at 52 weeks in individuals with trochanteric fractures. Secondary outcomes include revision surgery rates, fracture healing rates, fracture related adverse events, and health-related quality of life, including the Parker mobility score and Harris Hip Score.

DETAILED DESCRIPTION:
Hip fractures are becoming a more prevalent issue worldwide, leading to profound morbidity, and in some cases, mortality. Currently the most common method of surgical treatment includes the use of a sliding hip screw over a Gamma intramedullary nail, but there is conflicting evidence regarding which device has a lower revision surgery rate and complication rate. Recent improvements in implant design of the Gamma3 nail, demonstrating decreased rates of femoral shaft fractures and improved function, provide compelling rationale for the conduct of a large, definitive trial.

This trial is a definitive, multi-center, concealed randomized controlled trial. Surgeons will use one of the two surgical strategies in patients who have sustained a trochanteric fracture; the Gamma3 intramedullary nail or the sliding hip screw. Clinical assessments will occur at the time of hospital admission, post-surgery, 13 weeks, 26 weeks, 52 weeks, and 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women aged 18 years and older (with no upper age limit).
2. An intertrochanteric fracture (stable or unstable), AO Type 31-A1 or 31-A2, confirmed with anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
3. Low energy fracture (defined as a fall from standing height).
4. No other major trauma.
5. Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
6. Anticipated medical optimization of the patient for operative fixation of the proximal femur.
7. Operative treatment within 7 days after the trauma.(Operative treatment should take place as soon as possible as permitted by each institution's standard of care.)
8. Provision of informed consent by patient or proxy.

Exclusion Criteria:

1. Associated major injuries of the lower extremity (i.e., ipsilateral and/or contralateral fractures of the foot, ankle, tibia, fibula, or knee; dislocations of the ankle, knee, or hip).
2. Retained hardware around the affected proximal femur.
3. Infection around the proximal femur (i.e., soft tissue or bone).
4. Patients with disorders of bone metabolism other than osteoporosis (i.e., Paget's disease, renal osteodystrophy, or osteomalacia).
5. Patients with Parkinson's disease severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation.
6. Patients with a subtrochanteric fracture.
7. Patients with a pathologic fracture.
8. Patients with a reverse oblique fracture pattern, fracture AO Type 31-A3.
9. Obesity in the judgment of the attending surgeon.
10. Off-label use of the implant.
11. Patients with a previous history of frank dementia that would interfere with assessment of the primary outcome (i.e., EQ-5D at 1 year).
12. Likely problems, in the judgment of the Site Investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.
13. Patient is enrolled in another ongoing drug or surgical intervention trial.
14. If the attending surgeon believes that there is another reason to exclude this patient from INSITE. This reason will be documented on the case report forms (CRFs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | Up to 104 weeks
  To assess the impact of Gamma3 intramedullary nails versus sliding hip screws on health-related quality of life as measured by the EuroQol-5D at 52 weeks in individuals with trochanteric fractures.

SECONDARY OUTCOMES:
Health Related Quality of Life | Up to 104 weeks
  To assess the impact of Gamma3 intramedullary nails versus sliding hip screws on health-related quality of life as measured with the Parker mobility score and the Harris Hip Score.
Fracture healing rates | Up to 104 weeks
  A fracture is to be considered healed when there is obliteration of the fracture lines by newly formed bone along the cortices and within the trabecular bone on anteroposterior and lateral (or oblique) radiographs.
Fracture-related adverse events | Up to 104 weeks
  Including mortality, femoral shaft fracture, avascular necrosis (although rare in trochanteric fractures), nonunion, malunion (shortening, varus deformity, valgus deformity and rotational malunion), implant breakage or failure, and infection (i.e., superficial and deep).
Revision surgery rates | Up to 104 weeks
  Any unplanned surgery after the initial fixation to promote fracture healing (non-union), relieve pain (avascular necrosis, early or late implant failure), treat infection, or improve function will be considered a study event.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, PhD, FRCSC, Principal Investigator — Global Research Solutions; Georgia Mitchell, Study Director — Stryker Trauma and Extremities
Locations (26):
- United States (7):
  - Community Regional Medical Center, Fresno, California
  - San Francisco General Hospital, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Scott&White Memorial Hospital, Temple, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- Canada (2):
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - St. Michael's Hospital, Toronto, Ontario
- China (3):
  - Chaoyang Hospital, Beijing, Beijing Municipality
  - Sixth People's Hospital, Shanghai, Shanghai Municipality
  - 2nd Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
- Colombia (2):
  - Clinica El Rosario Sede El Tesoro, Medellín, Antioquia
  - Hospital Universitario Santa Clara, Bogotá, Cundinamarca
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Robert-Bosch-Krankenhaus, Stuttgart
- Tsukuba Medical Center, Tsukuba, Ibaraki, Japan
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands
- Helse Sunnmore Alesund Sjukehus, Ålesund, Norway
- Charlotte Maxeke Johannesburg Academic Hospital, Parktown, South Africa
- United Kingdom (4):
  - Frenchay Hospital, Bristol
  - The Royal Liverpool University Hospital, Liverpool
  - The Royal Berkshire Hospital, Reading
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahrengart L, Tornkvist H, Fornander P, Thorngren KG, Pasanen L, Wahlstrom P, Honkonen S, Lindgren U. A randomized study of the compression hip screw and Gamma nail in 426 fractures. Clin Orthop Relat Res. 2002 Aug;(401):209-22. doi: 10.1097/00003086-200208000-00024. PMID 12151898
- [Background] Bhandari M, Schemitsch E, Jonsson A, Zlowodzki M, Haidukewych GJ. Gamma nails revisited: gamma nails versus compression hip screws in the management of intertrochanteric fractures of the hip: a meta-analysis. J Orthop Trauma. 2009 Jul;23(6):460-4. doi: 10.1097/BOT.0b013e318162f67f. PMID 19550235
- [Background] Parker MJ, Handoll HH. Gamma and other cephalocondylic intramedullary nails versus extramedullary implants for extracapsular hip fractures in adults. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD000093. doi: 10.1002/14651858.CD000093.pub4. PMID 18646058
- [Derived] Schemitsch EH, Nowak LL, Schulz AP, Brink O, Poolman RW, Mehta S, Stengel D, Zhang CQ, Martinez S, Kinner B, Chesser TJS, Bhandari M; INSITE Investigators. Intramedullary Nailing vs Sliding Hip Screw in Trochanteric Fracture Management: The INSITE Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317164. doi: 10.1001/jamanetworkopen.2023.17164. PMID 37278998